CLINICAL TRIAL: NCT02785016
Title: Prospective, Non-Randomized, Observational Trial of the Surgical Management for Suburethral Slings in Women With Stress Urinary Incontinence
Brief Title: Surgical Management for Suburethral Slings
Status: Recruiting | Type: Observational
Sponsor: Cantonal Hospital, Frauenfeld (Other)
Responsible Party: Principal Investigator, Prof. Dr. Volker Viereck, Prof. Dr., Cantonal Hospital, Frauenfeld
Other Study IDs: TVT 3D
Record Dates: First submitted 2016-05-19; First posted 2016-05-27 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress Urinary Incontinence; Suburethral Sling
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Stress Urinary Incontinence: Females with stress urinary incontinence, who undergo a tension free surgical sling procedure.

SUMMARY:
This is a prospective, non-randomized, observational, single center study in which subjects that have surgically-correctable Stress Urinary Incontinence undergo a suburethral sling operative procedure.

DETAILED DESCRIPTION:
The study will collect preoperative urologic testing, medical history, and subject quality of life patient questionnaires. Intraoperative procedural data will be collected.

Postoperative complications, urologic, testing, and subject questionnaires will be collected at intervals. The anatomic position of the device will be characterize by introital ultrasound testing.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has objective demonstrable signs of stress urinary incontinence (SUI), including patients with intrinsic sphincter deficiency (ISD). Objective testing includes: standing stress test, urodynamics evaluation, or pad test.
2. Patient is age 18 or older.
3. Patient agrees to participate in the study, including completion of all study-related procedures and evaluations, and documents this agreement by signing the IRB/EC-approved informed consent.
4. Patient is able to fill in all questionnaires (on judgement of investigator)

Exclusion Criteria:

1. Patient has an associated or suspected neurological disease.
2. Patient has an active lesion or present injury to perineum or urethra.
3. Patient has a urethral obstruction.
4. Patient has significant pelvic organ prolapse (Grade III/IV) requiring surgical treatment.
5. The subject has current urinary tract infection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects that have surgically-correctable Stress Urinary Incontinence and undergo a suburethral sling operative procedure.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Cure/improvement rate | 3 months
  Patients are classified as cured if the postoperative cough test (see Outcome 4 below) is negative and the degree of subjective suffering (see Outcome 2 below) improves to over 90% (VAS score of 0 or 1). Criteria for improvement are involuntary loss of only a few drops of urine during straining and an improvement of the degree of suffering to over 75% (VAS score of 2 or 3). All other patients are classified as therapeutic failures (even if they show marked improvement of one of the parameters compared with their preoperative status).

SECONDARY OUTCOMES:
Subjective symptom assessment by visual analogue scale | 3 and 6 months
  Scale: 0-10 (0-no suffering, 10-severe suffering)
Post-Operative Pain Assessment | 1 day
  Scale: 0-10 (0-no pain, 10-severe pain)
Standing Cough Stress Test | baseline, 3 and 6 months
  3 categories: negative/severe, if flow of urine is observed. negative/mild, if the loss of only a few drops is observed. positive, if no urine loss occurs.
King Health Questionnaire | pre-operation, 3 and 6 months
International Consultation on Incontinence Questionnaire | pre-operation, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Volker Viereck, Physican, Principal Investigator — Cantonal Hospital, Frauenfeld
Locations (1):
- Blasenzentrum, Cantonal Hospital, Frauenfeld, Thurgau, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided